CLINICAL TRIAL: NCT01575977
Title: Stress Analysis of Hip Dysplasia After Corrective Surgery
Brief Title: Stress Analysis of Hip Dysplasia
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Andrew Anderson, Associate Professor, University of Utah
Other Study IDs: 43600
Record Dates: First submitted 2012-03-06; First posted 2012-04-12 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study is to predict cartilage contact pressures in the hip after periacetabular osteotomy (PAO).

DETAILED DESCRIPTION:
PAO was designed as a joint preserving surgical procedure to compensate for a shallow acetabulum by re-orienting the acetabulum into a position that provides better coverage of the femoral head. Although the overall theory that increasing load bearing area (improving coverage of the femoral head) results in reduced joint stress is intuitive, the complex bony surface may not behave in this manner. It is possible that joint stress may increase when the acetabulum is reoriented into a position that increases load bearing area if post-operative joint congruency is worse than pre-operative.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 years
* Patients who have undergone periacetabular osteotomy by Dr. Peters for treatment of hip dysplasia.
* Patients who have previously participated in IRB #10983 "Comparative Stress Analysis of Hip Dysplasia".

Exclusion Criteria:

* Persons with a history of allergies to lidocaine or seafood.
* Children under the age of 18.
* Persons incarcerated, on trial, or parole.
* Women who are pregnant.
* Subjects who do not have high quality pre-operative images available or have not been surgically treated by periacetabular osteotomy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 18-40 years old
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
To predict cartilage contact pressures in the hip joint during simulated daily activities before and after periacetabular osteotomy (PAO) for correction of traditional dysplasia/retroversion. | 1 year post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Anderson, Principal Investigator — Orthopedic Surgery Operations